CLINICAL TRIAL: NCT02990442
Title: The Effect of Rapid Transcranial Magnetic Stimulation (rTMS) on Aggression in Forensic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Gary Chaimowitz, Head of Forensics, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1938
Record Dates: First submitted 2016-11-23; First posted 2016-12-13 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Aggression
Keywords: rTMS; Repetitive Transcranial Magnetic Stimulation; Brain Stimulation
MeSH Terms: conditions — Aggression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rTMS (Experimental): treatment with repetitive transcranial magnetic stimulation for 30 days
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — repetitive transcranial magnetic stimulation, 1Hz protocol to right dorsolateral pre frontal cortex (R_DLPFC)

SUMMARY:
Forensic patients will undergo 30 rTMS treatments, once per day each business day using a 1Hz frequency at the right dorso-lateral pre frontal cortex, located using modified BEAM F3. Patients will be assessed before and after the study with a battery of assessments and using 2 computer tasks: a ball passing task, and the Point Subtraction Aggression Paradigm (PSAP). The investigators will also monitor and record aggressive incidents that take place on the unit.

ELIGIBILITY:
Inclusion Criteria:

1. are voluntary and competent to consent to treatment
2. are a current Forensics inpatient at St. Joseph's West 5th Campus
3. demonstrate aggressive behavior as confirmed by a psychologist or psychiatrist including verbal and physical aggression
4. are between the ages of 18 and 65
5. have had no changes in dose or initiation of any psychotropic medication in the 4 weeks prior to motor threshold
6. are willing and able to adhere to the treatment schedule
7. pass the TMS adult Safety-Screening (TASS) Questionnaire

Exclusion Criteria:

1. Withdraw consent to participate in the study
2. fail the TASS Safety Screening Questionnaire
3. have a concomitant major unstable medical illness, cardiac pacemaker or implanted medication pump, or a significant history of seizures
4. have active suicidal intent
5. are pregnant as confirmed by pregnancy test completed as part of pre-study screening
6. have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any significant history of seizure except those therapeutically induced by electroconvulsive therapy (ECT), cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis
7. have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
8. currently (or in the last 4 weeks) take more than lorazepam 2 mg daily (or equivalent) due to seizure risk or any dose of an anticonvulsant due to the potential to limit rTMS efficacy
9. non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Change in Aggressive Incident Scale (AIS) | 30 days
  ranking scale of aggressive incidents

OTHER OUTCOMES:
Change in Ball sharing task score | 30 days
  computer task
Change in Point Subtraction Aggression Paradigm (PSAP) | 30 days
  computer task

CONTACTS AND LOCATIONS:
Overall Officials: Gary Chaimowitz, MD, FRCPC, Principal Investigator — Head of Forensics
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No